CLINICAL TRIAL: NCT01712412
Title: Phase 2a Study of IW-9179 to Treat Functional Dyspepsia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-112-201
Record Dates: First submitted 2012-10-11; First posted 2012-10-23 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2013-07

CONDITIONS: Dyspepsia; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IW-9179 (Experimental): Oral IW-9179 taken daily for two weeks
  Interventions: Drug: IW-9179
- Placebo (Placebo Comparator): Oral placebo taken daily for two weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IW-9179
  Arms: IW-9179
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this study are to determine the safety and efficacy of IW-9179 administered to patients with functional dyspepsia (FD).

ELIGIBILITY:
Inclusion Criteria:

* Patient meets ROME III criteria for functional dyspepsia (FD)
* Patient has a normal esophagogastroduodenoscopy (EGD) either during the Screening Period or within 2 years of the Screening Visit
* Patients who EITHER:

  1. Have not used a proton pump inhibitor (PPI) within 4 weeks of the Screening Visit, OR
  2. Have used a PPI at a stable dose for at least 4 weeks prior to the Screening Visit;
* Patient meets symptom severity criteria in the Pretreatment Period
* Patient is fluent and literate in Dutch, French, or English

Exclusion Criteria:

* Patient meets criteria for gastroesophageal reflux disease (GERD, stable regimen of PPIs acceptable), constipation, diarrhea, lower abdominal pain, or gastroparesis
* Patient has a history of inflammatory bowel disease, chronic pancreatitis, small intestinal bacterial overgrowth, celiac disease, lactose intolerance, polycystic kidney disease, interstitial cystitis, or scleroderma
* Any significant neurological disease or a history of cancer (resected basal cell or squamous cell carcinoma of the skin is acceptable; complete remission of other cancers for 5 years or longer is also acceptable)
* History of active alcoholism or drug addiction within 12 months prior to the Screening Visit
* Hospitalized for a psychiatric condition or has made a suicide attempt during the two years before the Screening Visit
* Any organic or structural disease that can cause abdominal pain or discomfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Rate of treatment-emergent adverse events | Reported at any time after the first dose, including the 14 days of treatment and 7 days of follow up
Change from baseline 12-lead electrocardiogram (ECG) at day 14 of treatment | Baseline values taken just prior to first dose (day 1) compared with values taken on the last day of treatment (day 14)
Change from baseline clinical laboratory evaluations at the last day of treatment (day 14) | Baseline values taken just prior to first dose (day 1) compared with values taken on the last day of treatment (day 14)
Change from baseline vital signs at the day 14 visit and at the end of the study (7 days after the last dose) | Baseline values taken prior to first dose (day 1) compared with values taken at the day 14 visit (14 days after first dose) and at the end of the study (21 days after the first dose)

SECONDARY OUTCOMES:
Post-meal Symptom Severity (PMSS) Assessment | Completed at day 1 and day 14 of the Treatment Period
  Assessments completed at 15 min prior to dose, just prior to dose, and every 15 minutes after the first dose through 240 minutes (4 hours after first dose)
Daily Patient Symptom Severity (PSS) Assessment | Average of daily assessments for the 2 weeks just prior to the first dose compared to: 1) the average of the 2 week treatment period, 2) the average of the first week of treatment and 3) the average of the second week of treatment
  Assessments recorded on a daily basis
Weekly Symptom Relief (SR) Assessments | Average of week 1 and week 2 prior to treatment compared with the week 1 and week 2 during treatment
  Assessments recorded on a weekly basis weekly
Nepean Dyspepsia Index | Baseline NDI score (collected just prior to first dose) compared with End of Treatment NDI (collected just prior to last dose)

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (7):
  - AZ Sint-Lucas Brugge, Bruges
  - Antwerp University Hospital, Edegem
  - Z.O.L. - Campus St. Jan, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Ambroise Pare, Mons
  - H. Hartziekenhuis Roselare-Menen vzw, Roeselare
- Netherlands (8):
  - FlevoResearch, Almere Stad
  - PreCare Trial and Recruitment, Beek
  - Andromed Breda, Breda
  - Andromed Eindhoven, Eindhoven
  - Andromed Noord, Groningen
  - Andromed Leiden, Leiden
  - Maastricht University Med Ctr, Maastricht
  - Andromed Rotterdam, Rotterdam